CLINICAL TRIAL: NCT03075072
Title: Hippocampal Sparing Whole Brain Radiation Versus Stereotactic Radiation (SRS) in Patients With 5-20 Brain Metastases: A Phase III, Randomized Clinical Trial
Brief Title: Hippocampal Sparing Whole Brain Radiation Versus Stereotactic Radiation in Patients With 5-20 Brain Metastases: A Phase III, Randomized Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ayal Aizer, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-305
Record Dates: First submitted 2017-03-01; First posted 2017-03-09 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Brain Metastases
Keywords: Brain metastases; Brain metastasis; Lung cancer; Melanoma; Breast cancer; Kidney cancer; Renal cell carcinoma; Stereotactic radiation; Stereotactic radiosurgery; SRS; Stereotactic; Whole brain radiation; WBRT; Hippocampal avoidance; Hippocampal sparing; Hippocampal; Hippocampus; Radiation; Quality of Life; Neurocognitive; Neurocognition; Survival; Salvage; MDASI; Chemotherapy; Recurrence
MeSH Terms: conditions — Brain Neoplasms; Lung Neoplasms; Melanoma; Breast Neoplasms; Kidney Neoplasms; Carcinoma, Renal Cell; Recurrence | interventions — Radiosurgery; Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Whole Brain Radiation (Active Comparator): * MRI will be performed prior to radiation is administered
  * A hippocampal sparing approach will be used when possible
  * Dose will be 30 Gy in 10 fractions
  Interventions: Radiation: Whole brain radiation
- Stereotactic Radiation (SRS) (Experimental): * MRI will be performed prior to radiation is administered
  * Radiation will be given in 1-5 fractions (dose depends on the size of the tumor that will be treated)
  Interventions: Radiation: Stereotactic radiation (SRS)

INTERVENTIONS:
Radiation: Whole brain radiation — Treatment of the whole brain with radiation. When possible the hippocampus will be spared from radiation.
  Arms: Whole Brain Radiation
Radiation: Stereotactic radiation (SRS) — Focused radiation to each individual brain metastasis without treatment of the remainder of the brain.
  Arms: Stereotactic Radiation (SRS)

SUMMARY:
This research study is studying two different types of radiation as treatment for brain metastases (tumors in the brain that spread from a cancer that originated elsewhere in the body)

DETAILED DESCRIPTION:
This research study is a Phase III clinical trial. Phase III clinical trials examine the safety and effectiveness of a treatment, often comparing it to another known treatment. In this case, the investigators are specifically looking at differences between two forms of radiation treatment in terms of subsequent quality of life.

In this research study, the investigators are comparing stereotactic (focused, pinpoint) radiation (in which each tumor is narrowly targeted) against whole brain radiation (radiation targeting the entire brain) in the treatment of brain metastases. Currently whole brain radiation is the standard option for patients with 5-20 brain metastases. Stereotactic radiation is the standard option for patients with 1-4 brain metastases. Among patients with 1-4 brain metastases, recently published studies suggest that stereotactic radiation results in fewer neurologic side effects than whole brain radiation. It also yields better quality of life in this population. It remains unknown whether stereotactic radiation improves quality of life in patients with 5-20 brain metastases relative to whole brain radiation. In this study, the investigators seek to determine which of the two methods of study treatment results in a better subsequent quality of life for patients with 5-20 brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a biopsy proven solid malignancy with untreated (by radiation) intracranial lesions radiographically consistent with or pathologically proven to be brain metastases. Patients who have undergone prior systemic therapy are eligible
* Five-twenty intracranial lesions must be present on MRI of the brain
* Age 18-80 years at diagnosis of brain metastases
* Karnofsky performance status of at least 70

Exclusion Criteria:

* Participants who have undergone prior radiation for brain metastases.
* Patients who have undergone resection of one or more brain metastases but who have not yet started adjuvant radiotherapy are eligible for the study
* Participants who cannot undergo a brain MRI
* Participants who cannot receive gadolinium (MRI contrast)
* Participants with stage IV-V chronic kidney disease or end stage renal disease
* Participants with widespread, definitive leptomeningeal disease
* Participants with small cell lung cancer, lymphoma, or myeloma
* Participants with a maximum tumor diameter exceeding 5 cm (if not resected)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2024-11-07 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Survey (symptoms and interference) | 6 months
  Questionnaire - MD Anderson Symptom Inventory - Brain Tumor (MDASI-BT)

SECONDARY OUTCOMES:
Overall survival | Through study completion, an average of 1 year
  Clinical Parameter
Neurologic survival | Through study completion, an average of 1 year
  Clinical parameter to be assessed via review of study visits and medical records indicating cause of death (neurologic versus systemic)
Incidence and time to detection of new brain metastases | Through study completion, an average of 1 year
  Radiographic assessment of first appearance of new brain metastases
Incidence and time to local recurrence of treated brain tumor(s) | Through study completion, an average of 1 year
  Radiographic assessment of first local recurrence in the 5-20 brain metastases that were initially treated with radiation
Incidence and time to development of radiation necrosis | Through study completion, an average of 1 year
  Radiographic assessment of first appearance of radiation necrosis
Incidence and time to development of leptomeningeal disease | Through study completion, an average of 1 year
  Radiographic assessment of first appearance of leptomeningeal disease
Incidence and time to salvage craniotomy | Through study completion, an average of 1 year
  Clinical assessment of first use of neurosurgical resection as salvage therapy
Incidence and time to additional radiotherapeutic treatments | Through study completion, an average of 1 year
  Clinical assessment of first use of salvage brain-directed radiation
Incidence and time to the development of seizures | Through study completion, an average of 1 year
  Clinical assessment of first post-treatment seizure as assessed during routine study visits and via medical record review
Incidence and time to neurocognitive decline | 1 year
  Scale
Performance status | Through study completion, an average of 1 year
  Questionnaire - Karnofsky performance status

CONTACTS AND LOCATIONS:
Overall Officials: Ayal Aizer, MD MHS, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No